CLINICAL TRIAL: NCT06935578
Title: RAre, But Not aLone: a Large Italian Network to Empower the Impervious diaGNostic Pathway of Rare cerEbrovascular Diseases (ALIGNED)
Acronym: ALIGNED
Status: Recruiting | Type: Observational
Sponsor: Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta (Other)
Responsible Party: Sponsor
Other Study IDs: ALIGNED
Record Dates: First submitted 2025-04-02; First posted 2025-04-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: CADASIL; CADASIL (Diagnosis); Moya Moya Disease; Moyamoya; Moyamoya Syndrome; Sneddon Syndrome; Fabry Disease; COL4A1\2
Keywords: Rare Cerebrovascular Diseases; italian network; CADASIL; COL4A1 syndrome; Fabry Disease; Sneddon Syndrome; Moyamoya arteriopathy; COL4A1/2
MeSH Terms: conditions — CADASIL; Disease; Moyamoya Disease; Sneddon Syndrome; Fabry Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Cerebrovascular diseases (CVDs) are one leading cause of morbidity and mortality worldwide. Despite intensive investigations, more than 30% of strokes remain of undetermined origin. Rare Cerebrovascular Diseases (rCVDs), including heritable (i.e., CADASIL, COL4A1 syndrome, Fabry disease) and acquired conditions (i.e., Sneddon syndrome, Moyamoya arteriopathy) account for a proportion of these strokes. However, rCVDs are often misdiagnosed since clinicians are not able to recognize them. Although rare, the identification of these stroke causes is important to establish appropriate management measures, including genetic counselling, and, if available, therapy. The lack of data on phenotype and clinical course of rCVDs, given the paucity of published series, makes the diagnosis and the development of therapies challenging. Furthermore, the molecular characterization of rCVDs is still lacking, despite progresses achieved in common stroke by applying high throughput approaches as multi-omics. Since the diagnosis and care of rCVDs require adequate expertise and instrumental tools, clinical and research activities are usually reserved to few specialized centers, mostly located in the North of Italy, leading patients to expensive trips for consultations. Therefore, the creation of a clinical and research network aimed at improving the diagnostic pathways of rCVDs is highly needed to improve the number of patients with rCVDs to better define the clinical phenotype and to transfer the knowledge on rCVDs in other centers overall Italy filling the geographical gap affecting Southern Italy.

ELIGIBILITY:
Inclusion Criteria:

* patients with a clinical, genetic and/or neuroradiological diagnosis of rCVD (CADASIL, Fabry's disease, COL4A1, Sneddon's syndrome or Moyamoya arteriopathy), who have had at least one brain MRI study;

Exclusion Criteria:

* na

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults, male and female patients affected by a Rare Cerebrovascular Disease (rCVD)
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Describe the phenotypic characteristics of rCVD patients | 0-12 months
  To describe the phenotypic characteristics of rCVD patients. All patients will complete a standardized neurological assessment consisting of anamnestic data collection (family history of neurological pathology, and in particular of rCVD, cardiovascular risk factors, medications taken, comorbidities, recent or previous head injuries) and a complete physical examination.
Assess the natural history of disease | 0-12 months
  To develop a new, unique, and large registry on rCVDs recruiting a large number of patients (500) , patients will be recruited by all the participating clinical centers

SECONDARY OUTCOMES:
Identify the molecular mechanisms | 12-30 months
  Identify the molecular mechanisms underlying rCVD, targeted/quantitative approaches will validate the emerged key molecular features (e.g by transcriptomic, proteomic, metabolomic, and lipidomic approaches).
Identify biomarkers | 12-30 months
  Identify reliable and usable circulating biomarkers for the diagnosis of rCVD by applying mass spectrometry-based cutting-edge technologies for an unbiased identification of differentially abundant candidates (e.g. proteins or metabolites), and for their validation and simultaneous assessment in multi-marker panels
Provide the best clinical and therapeutic management | 12-30 months
  Implement the virtual multi-specialty and multicenter rCVD case-sharing model in order to provide the best clinical and therapeutic management of the patients taken in. A team of specialists with expertise in each rCVD, comprising neurologists, neurosurgeons, neuro-radiologists, interventional radiologists, neuropsychiatrists, geneticists, neurophysiologists and/or psychologists, will schedule virtual monthly meetings to discuss the diagnosis and provide individual patients with the best diagnostic and management paths. A specific platform for second opinion consultations will be created by using the existing telemedicine platform.

CONTACTS AND LOCATIONS:
Locations (17):
- Italy (17):
  - Ospedale Regionale Generale "F. Miulli", Acquaviva delle Fonti, Acquaviva delle Fonti, BA
  - ASST Melegnano Martesana, Melegnano, MI
  - Neurologia Stroke Unit dell'Asst Rhodense, Rho, Mi
  - Fondazione Istituto G. Giglio, Cefalù, Cefalù, PA
  - UO Neurologia degli Ospedali di Cesena e Forlì, Ospedale Bufalini Cesena ed Ospedale Morgagni-Pierantoni (Ausl della Romagna), Cesena
  - ASST di Cremona, Cremona
  - Ospedale "Spaziani" di Frosinone, Frosinone
  - U.O. Neurologia, Ospedale Sant'Andrea, La Spezia, La Spezia
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - Fondazione IRCCS Istituto Neurologico Carlo Besta, Milan
  - Ospedale Luigi Sacco, ASST Fatebenefratelli Sacco, Milan
  - Stroke Unit Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico di Milano, Milan
  - IRCCS Policlinico San Matteo, Pavia, Pavia
  - Neurologia d'Urgenza e Stroke Unit dell'Ospedale di Pescara, Pescara
  - Neurologia dell'Ospedale Sandro Pertini - ASL Roma2, Roma
  - Policlinico Tor Vergata, UOSD Stroke Unit, Roma
  - Neurologia PO Levante Asl 2 Savonese, Savona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Caponnetto V, Ornello R, De Matteis E, Papavero SC, Fracasso A, Di Vito G, Lancia L, Ferrara FM, Sacco S. The COVID-19 Pandemic as an Opportunity to Improve Health Care Through a Nurse-Coordinated Multidisciplinary Model in a Headache Specialist Center: The Implementation of a Telemedicine Protocol. Telemed J E Health. 2022 Jul;28(7):1016-1022. doi: 10.1089/tmj.2021.0414. Epub 2021 Nov 9. PMID 34756108
- [Background] Banfi C, Baetta R, Barbieri SS, Brioschi M, Guarino A, Ghilardi S, Sandrini L, Eligini S, Polvani G, Bergman O, Eriksson P, Tremoli E. Prenylcysteine oxidase 1, an emerging player in atherosclerosis. Commun Biol. 2021 Sep 21;4(1):1109. doi: 10.1038/s42003-021-02630-z. PMID 34548610
- [Background] Degan D, Ornello R, Tiseo C, De Santis F, Pistoia F, Carolei A, Sacco S. Epidemiology of Transient Ischemic Attacks Using Time- or Tissue-Based Definitions: A Population-Based Study. Stroke. 2017 Mar;48(3):530-536. doi: 10.1161/STROKEAHA.116.015417. Epub 2017 Jan 31. PMID 28143922
- [Background] Sacco S, Marini C, Toni D, Olivieri L, Carolei A. Incidence and 10-year survival of intracerebral hemorrhage in a population-based registry. Stroke. 2009 Feb;40(2):394-9. doi: 10.1161/STROKEAHA.108.523209. Epub 2008 Nov 26. PMID 19038914
- [Background] Romani I, Nencini P, Sarti C, Pracucci G, Zedde M, Nucera A, Cianci V, Moller J, Toni D, Orsucci D, Casella C, Pinto V, Palumbo P, Barbarini L, Bella R, Ragno M, Scoditti U, Mezzapesa DM, Tassi R, Diomedi M, Cavallini A, Volpi G, Chiti A, Bigliardi G, Sacco S, Linoli G, Ricci S, Giordano A, Bonetti B, Rasura M, Cecconi E, Princiotta Cariddi L, Curro Dossi R, Melis M, Consoli D, Guidetti D, Biagini S, Accavone D, Inzitari D. Fabry-Stroke Italian Registry (FSIR): a nationwide, prospective, observational study about incidence and characteristics of Fabry-related stroke in young-adults. Presentation of the study protocol. Neurol Sci. 2022 Apr;43(4):2433-2439. doi: 10.1007/s10072-021-05615-2. Epub 2021 Oct 5. PMID 34609660
- [Background] Bersano A, Markus HS, Quaglini S, Arbustini E, Lanfranconi S, Micieli G, Boncoraglio GB, Taroni F, Gellera C, Baratta S, Penco S, Mosca L, Grasso M, Carrera P, Ferrari M, Cereda C, Grieco G, Corti S, Ronchi D, Bassi MT, Obici L, Parati EA, Pezzini A, De Lodovici ML, Verrengia EP, Bono G, Mazucchelli F, Zarcone D, Calloni MV, Perrone P, Bordo BM, Colombo A, Padovani A, Cavallini A, Beretta S, Ferrarese C, Motto C, Agostoni E, Molini G, Sasanelli F, Corato M, Marcheselli S, Sessa M, Comi G, Checcarelli N, Guidotti M, Uccellini D, Capitani E, Tancredi L, Arnaboldi M, Incorvaia B, Tadeo CS, Fusi L, Grampa G, Merlini G, Trobia N, Comi GP, Braga M, Vitali P, Baron P, Grond-Ginsbach C, Candelise L; Lombardia GENS Group*. Clinical Pregenetic Screening for Stroke Monogenic Diseases: Results From Lombardia GENS Registry. Stroke. 2016 Jul;47(7):1702-9. doi: 10.1161/STROKEAHA.115.012281. Epub 2016 May 31. PMID 27245348
- [Background] Bersano A, Bedini G, Markus HS, Vitali P, Colli-Tibaldi E, Taroni F, Gellera C, Baratta S, Mosca L, Carrera P, Ferrari M, Cereda C, Grieco G, Lanfranconi S, Mazucchelli F, Zarcone D, De Lodovici ML, Bono G, Boncoraglio GB, Parati EA, Calloni MV, Perrone P, Bordo BM, Motto C, Agostoni E, Pezzini A, Padovani A, Micieli G, Cavallini A, Molini G, Sasanelli F, Sessa M, Comi G, Checcarelli N, Carmerlingo M, Corato M, Marcheselli S, Fusi L, Grampa G, Uccellini D, Beretta S, Ferrarese C, Incorvaia B, Tadeo CS, Adobbati L, Silani V, Farago G, Trobia N, Grond-Ginsbach C, Candelise L; Lombardia GENS-group. The role of clinical and neuroimaging features in the diagnosis of CADASIL. J Neurol. 2018 Dec;265(12):2934-2943. doi: 10.1007/s00415-018-9072-8. Epub 2018 Oct 11. PMID 30311053
- [Background] Bersano A, Bedini G, Nava S, Acerbi F, Sebastiano DR, Binelli S, Franceschetti S, Farago G, Grisoli M, Gioppo A, Ferroli P, Bruzzone MG, Riva D, Ciceri E, Pantaleoni C, Saletti V, Esposito S, Nardocci N, Zibordi F, Caputi L, Marzoli SB, Zedde ML, Pavanello M, Raso A, Capra V, Pantoni L, Sarti C, Pezzini A, Caria F, Dell' Acqua ML, Zini A, Baracchini C, Farina F, Sanguigni S, De Lodovici ML, Bono G, Capone F, Di Lazzaro V, Lanfranconi S, Toscano M, Di Piero V, Sacco S, Carolei A, Toni D, Paciaroni M, Caso V, Perrone P, Calloni MV, Romani A, Cenzato M, Fratianni A, Ciusani E, Prontera P, Lasserve ET, Blecharz K, Vajkoczy P, Parati EA; GEN-O-MA study group. GEN-O-MA project: an Italian network studying clinical course and pathogenic pathways of moyamoya disease-study protocol and preliminary results. Neurol Sci. 2019 Mar;40(3):561-570. doi: 10.1007/s10072-018-3664-z. Epub 2019 Jan 3. PMID 30604336
- [Background] Bersano A, Morbin M, Ciceri E, Bedini G, Berlit P, Herold M, Saccucci S, Fugnanesi V, Nordmeyer H, Farago G, Savoiardo M, Taroni F, Carriero M, Boncoraglio Giorgio B, Perucca L, Caputi L, Parati Eugenio A, Kraemer M. The diagnostic challenge of Divry van Bogaert and Sneddon Syndrome: Report of three cases and literature review. J Neurol Sci. 2016 May 15;364:77-83. doi: 10.1016/j.jns.2016.03.011. Epub 2016 Mar 5. PMID 27084221
- [Background] Panara V, Navarra R, Mattei PA, Piccirilli E, Bartoletti V, Uncini A, Caulo M. Correlations between cervical spinal cord magnetic resonance diffusion tensor and diffusion kurtosis imaging metrics and motor performance in patients with chronic ischemic brain lesions of the corticospinal tract. Neuroradiology. 2019 Feb;61(2):175-182. doi: 10.1007/s00234-018-2139-5. Epub 2018 Dec 5. PMID 30519889